CLINICAL TRIAL: NCT00725270
Title: Treatment of Schizoaffective Disorder Using Mifepristone
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Stanford University (Other)
Collaborators: Pritzker Family Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-06012008-1191; 76458
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Psychotic Disorders; Depressive Disorder, Major; Depressive Disorder
MeSH Terms: conditions — Psychotic Disorders; Depressive Disorder, Major; Depressive Disorder | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Patients will be randomized to placebo
  Interventions: Drug: Placebo Oral Tablet
- Mifepristone (Experimental): Patients will be randomized to mifepristone
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — 600 mg of mifepristone
  Arms: Mifepristone
Drug: Placebo Oral Tablet — Placebo comparator
  Arms: Placebo

SUMMARY:
This study tests the hypothesis that mifepristone will diminish cognitive distortion and alleviate psychosis in patients with schizoaffective disorder.

DETAILED DESCRIPTION:
You are invited to participate in a research study which evaluates the effectiveness of mifepristone (RU 486) in rapidly reducing the symptoms associated with schizoaffective disorder. Our group believes that the cognitive deficits (a decline in the ability to think clearly) and psychosis (hallucinations or delusions) exhibited in some affective disorders are driven by an excess of stress hormone effects (hypercortisolemia). Often the origin of this hormonal imbalance is unknown. Current treatment for schizoaffective disorder (characterized by mood swings and hallucinations and/or delusions) involves using a combination of antidepressant medication (for mood elevation), mood stabilizing medications (to prevent extreme high and low moods) and antipsychotic medication (for the correction of altered thinking). While these therapies are often effective, they can take several weeks or longer to work. We hope to uncover a quick, effective, safe therapy for the treatment of individuals with your condition.

ELIGIBILITY:
Inclusion Criteria:The subjects will be 30 inpatients or outpatients with schizoaffective disorder. Exclusion Criteria:Subjects must be between the ages of eighteen and seventy-five without major medical problems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1998-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keller, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Cherian K, Schatzberg AF, Keller J. HPA axis in psychotic major depression and schizophrenia spectrum disorders: Cortisol, clinical symptomatology, and cognition. Schizophr Res. 2019 Nov;213:72-79. doi: 10.1016/j.schres.2019.07.003. Epub 2019 Jul 12. PMID 31307859

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Mifepristone
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mifepristone | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (15.9) | 27.29 (8.6) | 31.08 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 7 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive Psychotic Symptoms Over the Course of Treatment
Description: Utilized the Positive Symptoms Subscale of the Brief Psychiatric Rating Scale is assess psychotic symptoms. Range for the subscale is 4-28, with 4 = no positive symptoms
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mifepristone
Number analyzed (Participants) | 5 | 7
units on a scale
  Baseline PSS Scores | 12.0 (5.2) | 7.57 (3.5)
  Day 9 PSS scores | 11.0 (6.4) | 6.0 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Mifepristone; Repeated Measures ANOVA was run on the Positive Symptom Scale of the Brief Psychiatric Rating Scale, using Baseline and Day 9 ratings. Below is the medication * time interaction; Test type: Superiority or Other; p = .812, Mixed Models Analysis

2. Primary Outcome: Change in Mood Symptoms
Description: Utilized the Hamilton Depression Rating Scale, 21-item version to assess depressive symptoms, with a range of 0-63, with higher scores indicating greater levels of depression.
Time Frame: Baseline and Day 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mifepristone
Number analyzed (Participants) | 5 | 7
units on a scale
  Baseline | 26.2 (10.3) | 24.86 (4.0)
  Day 9 | 19.0 (8.3) | 13.57 (5.5)
Statistical Analysis 1: Comparison: Placebo vs Mifepristone; Test type: Superiority or Other; p = .203, Mixed Models Analysis; eta sq = .157

ADVERSE EVENTS:
Arm/Group | Placebo | Mifepristone
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No